CLINICAL TRIAL: NCT04493060
Title: Phase II Study of Niraparib and TSR-042 in Patients With Germline or Somatic BRCA1/2 and PALB2-Related Pancreatic Cancer
Brief Title: Niraparib and Dostarlimab for the Treatment of Germline or Somatic BRCA1/2 and PALB2 Mutated Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1841; NCI-2020-05352 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1841 (Other: Mayo Clinic in Rochester); 18-003525 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — dostarlimab; Immunoglobulin G; Disulfides; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (niraparib, dostarlimab) (Experimental): Patients receive niraparib PO QD on days 1-21. Patients also receive dostarlimab IV over 30 minutes on day 1 Q3W for cycles 1-4 and Q6W for subsequent cycles. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dostarlimab; Drug: Niraparib

INTERVENTIONS:
Biological: Dostarlimab — Given IV
  Other Names: ANB011; Immunoglobulin G4, Anti-programmed Cell Death Protein 1 (PDCD1) (Humanized Clone ABT1 Gamma4-chain), Disulfide with Humanized Clone ABT1 Kappa-chain, Dimer; TSR 042; TSR-042; TSR042
Drug: Niraparib — Given PO
  Other Names: MK-4827; MK4827

SUMMARY:
This phase II trial studies how well niraparib and dostarlimab work in treating patients with germline or somatic BRCA1/2 and PALB2 mutated pancreatic cancer that has spread to other places in the body (metastatic). Niraparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as dostarlimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving niraparib and dostarlimab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine antitumor activity as measured by disease control rate at 12 weeks (DCR12) as assessed using immune-modified Response Evaluation Criteria in Solid Tumors (iRECIST) in select homologous recombination repair (HRR) deficient pancreatic cancer patients with HRR deficiency (defined as mutations in BRCA 1/ 2, or PALB2).

SECONDARY OBJECTIVES:

I. To assess adverse events according to the current National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) and other safety parameters.

II. To assess the time to next treatment (TTNT), objective response rate (ORR), time to and duration of response and duration of confirmed stable disease according to iRECIST.

III. To assess progression-free survival. IV. To assess overall survival.

CORRELATIVE RESEARCH OBJECTIVES:

I. To assess germline deoxyribonucleic acid (DNA) and serum markers of immune response.

II. To determine changes in circulating tumor DNA (ctDNA) profile after therapy with a PARP inhibitor (i) and a PD-1 inhibitor.

III. To study mechanisms of resistance in ctDNA profile after therapy with a PARPi and a PD-1 inhibitor.

IV. To assess the tumor microenvironment for immune related changes (immune infiltration, PD-L1 and PD-1 expression, tumor-infiltrating lymphocytes [TIL]).

V. To assess genetic profile of the tumor pre- and post-treatment. VI. To determine changes in the cytokine profile pre- and post-treatment.

OUTLINE:

Patients receive niraparib orally (PO) once daily (QD) on days 1-21. Patients also receive dostarlimab intravenously (IV) over 30 minutes on day 1 every 3 weeks (Q3W) for cycles 1-4 and every 6 weeks (Q6W) for subsequent cycles. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months until progressive disease (PD), and then every 6 months for up to 5 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Presence of either a germline deleterious mutation or somatic deleterious mutation in any one of the genes in our proposed gene-panel as determined by any of the commercially available or institutional testing platforms. Note: The somatic mutation could be either on a tissue-based test or the circulating tumor DNA (ctDNA)-based assay. The 6 genes that would determine eligibility would be: BRCA1/2, PALB2, BARD1, RAD51c, RAD51d
* Provide written informed consent
* Histological/cytological confirmation of diagnosis of metastatic pancreatic ductal adenocarcinoma
* At least one but no more than two prior lines of systemic therapy for metastatic disease (maintenance therapy is not considered a line of treatment)

  * Note: Patients who have not had any prior chemotherapy can refuse chemotherapy and be considered eligible. This refusal and their reason for refusal would have to be documented
* Received a platinum agent as part of first or second line treatment (unless contraindicated)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or estimated glomerular filtration rate (eGFR) >= 60 mL/min using the Cockcroft-Gault Equation (=< 14 days prior to registration)
* Hemoglobin >= 9.0 g/dL (=< 14 days prior to registration)
* Absolute neutrophil count >= 1500/uL (=< 14 days prior to registration:)
* Platelets >= 100 x 10^9/L (=< 14 days prior to registration)
* Total bilirubin =< 1.5 x ULN, (2.0 x ULN for subjects with Gilbert's disease) (=< 14 days prior to registration:)
* Aspartate transaminase (AST) and alanine transaminase (ALT) =< 2.5 x ULN (for subjects with hepatic metastases =< 5 x ULN) (=< 14 days prior to registration). Note: One time repeat testing to meet eligibility is allowed. If more testing is required, discuss with principal investigator (PI)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants. Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (=< 14 days prior to registration)
* Evaluable or measurable disease per iRECIST
* Life expectancy of >= 3 months
* Willingness to consent to translational studies
* Willingness to undergo repeat biopsies of tumor lesions amenable to biopsy

  * Note: While biopsies are mandatory, subjects are allowed to participate if no lesions are amenable to biopsy, or if biopsy is not possible due to safety
* Willingness to not donate blood during the study or for 90 days after the last dose of study treatment
* Willingness to not breastfeed during the study or for 90 days after the last dose of study treatment
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

Exclusion Criteria:

* Known hypersensitivity to any component of study treatments (either niraparib and/or TSR-042 or similar medications)
* Prior treatment with the combination of PARP inhibition and immunotherapy (either CTLA-4 or anti-PD1/PD-L1 therapies). Prior treatment consisting of monotherapy with either PARP inhibitors and/or with immunotherapy are allowed. Treatment with PARPi or PD1 inhibitor as the most recent treatment prior to enrollment is not allowed
* Patient experienced >= grade 3 immune-related adverse events (AE) with prior immunotherapy, with the exception of non-clinically significant lab abnormalities
* Radiotherapy =< 2 weeks prior to first study treatment or radionuclide treatment =< 4 weeks of first study treatment
* Live attenuated vaccine administration within 30 days prior to registration and/or expected during study period
* Known brain metastases, uncontrolled seizure disorder, or active neurologic disease which in the opinion of the investigator would impede participation within the trial. Subjects with treated brain metastases are allowed to enroll
* Allogeneic bone marrow transplantation or high-dose chemotherapy requiring hematopoietic stem cell rescue
* Received a transfusion (platelets or red blood cells) =< 4 weeks prior to registration

  * NOTE: patients are also deemed ineligible if they have received a transfusion =< 4 weeks prior to first dose of niraparib
* Received colony-stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) =< 4 weeks prior to registration

  * NOTE: patients are also deemed ineligible if they have received colony-stimulating factors =< 4 weeks prior to first dose of niraparib
* Known grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment
* Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* =< 4 weeks since receiving treatment with another investigational drug, or anti-cancer therapy, or within a time interval less than at least 5 half-lives of the investigational agent (whichever is shorter), or insufficient recovery (to the judgement of the investigator) from adverse events due to such a previously administered agent, except for alopecia prior to initiating protocol therapy. Bisphosphonate therapy and receptor activator of nuclear factor kappa-Β ligand (RANKL) inhibitors are not considered anti-cancer therapy
* Inadequate recovery from toxicity and/or complications from previous interventions, including due to major surgery to the judgement of the investigator. Minor surgery allowed up to 3 weeks from registration
* Primary or secondary immunodeficiency, including immunosuppressive disease, and immunosuppressive doses of corticosteroids (e.g., prednisone > 20 mg per day during 2 weeks prior to first study treatment) or other immunosuppressive medications at dose levels that to the judgement of the investigator would preclude participation within the past 4 weeks prior to registration. Subjects with human immunodeficiency virus (HIV) who are stable on highly active antiretroviral therapy (HAART) will not be excluded
* Participant has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected)
* Pregnant or lactating
* Clinically significant, active, bacterial infections that, to the judgement of the investigator makes it undesirable for the subject to participate in the study
* Persons of childbearing potential (POCBP) or those capable of causing pregnancy whose sexual partners are POCBP who are unwilling or unable to use an effective method of contraception for at least 1 month prior to study entry, for the duration of the study, and for at least 180 days after the last dose of study drug. Non-childbearing potential is defined as follows (by other than medical reasons):

  * >= 45 years of age and has not had menses for > 1 year
  * Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use an adequate barrier method throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient
* History or active TB (Bacillus tuberculosis) that in the investigators opinion would preclude participation within the study
* Any gastro-intestinal conditions that to the judgement of the investigator would interfere with the absorption of niraparib
* Active, known or suspected unstable auto-immune disease, are excluded from this study. Exceptions to this criterion are all auto-immune disease that have remained stable within the past 3 months on corticosteroids (=< prednisone 20 mg or equivalent) prior to first study treatment are allowed to enroll. Patients with autoimmune diseases that do not require active immunosuppression are also allowed to enroll

  * Note: Paraneoplastic disease as a cause of auto-immune phenomenon will not be considered as auto-immune disease and are allowed to enroll
* Evidence of serious uncontrolled medical disorder, active infection or mental disorder that, to the judgement of the investigator, makes it undesirable for the subject to participate in the study or that would jeopardize compliance with the protocol. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
* Prior malignancy which required active systemic treatment within 2 years prior to first study treatment. Exceptions are: successfully treated squamous cell carcinoma of the skin, superficial bladder cancer, and in situ carcinoma of the cervix. Since patients with BRCA 1/2 or PALB2 can have other tumors, as long as they have been definitively treated, it would not be considered an exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2025-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert R. McWilliams, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Niraparib, Dostarlimab): Patients receive niraparib PO QD on days 1-21. Patients also receive dostarlimab IV over 30 minutes on day 1 Q3W for cycles 1-4 and Q6W for subsequent cycles. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.>> >> Dostarlimab: Given IV>>
  >> Niraparib: Given PO
Period: Overall Study
Arm/Group | Treatment (Niraparib, Dostarlimab)
Started | 22
Completed | 18
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Niraparib, Dostarlimab)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Number of Prior Treatment(s) [Count of Participants; unit: Participants]
  1 | 3
  2 | 7
  3+ | 8
Mismatch Repair Status [Count of Participants; unit: Participants] — Population: One patient did not give information on mismatch repair status
  Participants
    Deficient: number analyzed (Participants) | 17
    Deficient | 2
    Proficient: number analyzed (Participants) | 17
    Proficient | 15
Deleterious Mutation [Count of Participants; unit: Participants]
  BRCA 1 | 5
  BRCA 2 | 12
  PALB2 | 1
Platinum Tx Exposure [Count of Participants; unit: Participants]
  Yes | 16
  No | 2
Refractory To Cancer Tx [Count of Participants; unit: Participants]
  Yes | 5
  No | 13

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate at 12 Weeks (DCR12)
Description: Will be assessed using the standard immune-modified Response Evaluation Criteria in Solid Tumors (iRECIST) criteria.
Time Frame: At 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Niraparib, Dostarlimab)
Number analyzed (Participants) | 18
Participants
  No Success | 13
  Success | 5

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The confirmed response rate (by iRECIST ) will be assessed.
Time Frame: Up to 4 years and 5 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Niraparib, Dostarlimab): Patients receive niraparib PO QD on days 1-21. Patients also receive dostarlimab IV over 30 minutes on day 1 Q3W for cycles 1-4 and Q6W for subsequent cycles. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  >
  >
  >
  >
  >
  > Dostarlimab: Given IV
  >
  >
  >
  >
  >
  > Niraparib: Given PO
Arm/Group | Treatment (Niraparib, Dostarlimab)
Number analyzed (Participants) | 18
Participants | 0

3. Secondary Outcome: Time to Next Treatment (TTNT)
Description: TTNT will be estimated using the Kaplan-Meier method.
Time Frame: From the end of study treatment to receiving the next treatment, assessed up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival (OS)
Description: OS will be estimated using the Kaplan-Meier method.
Time Frame: From study entry to death from any cause, assessed up to 4 years and 5 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment (Niraparib, Dostarlimab): Patients receive niraparib PO QD on days 1-21. Patients also receive dostarlimab IV over 30 minutes on day 1 Q3W for cycles 1-4 and Q6W for subsequent cycles. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  >>
  >> Dostarlimab: Given IV
  >>
  >> Niraparib: Given PO
Arm/Group | Treatment (Niraparib, Dostarlimab)
Number analyzed (Participants) | 18
months | 27.9 [27.3 to NA] — Not enough events to calculate upper bound

5. Secondary Outcome: Time to and Duration of Confirmed Response
Description: Will be assessed using the Kaplan-Meier method.
Time Frame: From the first documented date of confirmed response (complete response [CR] or partial response [PR]) to the date at which progression is first documented, assessed up to 5 years
Population: Since 0 responses, Time to and duration of confirmed response is Not Applicable. We didn't have a single confirmed response.
Groups:
- Treatment (Niraparib, Dostarlimab): Patients receive niraparib PO QD on days 1-21. Patients also receive dostarlimab IV over 30 minutes on day 1 Q3W for cycles 1-4 and Q6W for subsequent cycles. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.> >>
  >
  >> Dostarlimab: Given IV>
  >>
  >
  >> Niraparib: Given PO
Arm/Group | Treatment (Niraparib, Dostarlimab)
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS will be estimated using the Kaplan-Meier method.
Time Frame: From study entry to the first of either disease progression or death from any cause, assessed up to 4 years and 5 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Niraparib, Dostarlimab)
Number analyzed (Participants) | 18
months | 16.4 [13.6 to NA] — Not enough events to calculate upper bound

7. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The frequency and percentage of grade 3+ adverse events will be estimated. Will also assess AEs at least possibly related to treatment as well.
Time Frame: Up to 4 years and 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Niraparib, Dostarlimab)
Number analyzed (Participants) | 18
Participants
  Any Grade 3 or Higher | 15
  Any Grade 4 or Higher | 3
  Grade 5 | 2
  Hematologic Grade 3 or Higher | 9
  Hematologic Grade 4 or Higher | 1
  Hematologic Grade 5 | 0
  Non-Hematologic Grade 3 or Higher | 12
  Non-Hematologic Grade 4 or Higher | 2
  Non-Hematologic Grade 5 | 2

8. Other Pre Specified Outcome: Germline Deoxyribonucleic Acid (DNA) and Serum Markers of Immune Response
Description: Due to the limited sample size, these analyses will be hypothesis generating and descriptive in nature. Descriptive statistics will be summarized and the blood and tissue marker data will be correlated with clinical endpoints (response, DCR12, duration of response, OS, PFS, adverse events, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, will use the Fisher's exact test. For marker data used to predict binary outcomes (i.e. response versus [vs]. no response), will use logistic regression models.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Changes in Circulating Tumor DNA (ctDNA) Profile After Therapy With a PARP Inhibitor (i) and a PD-1 Inhibitor
Description: Due to the limited sample size, these analyses will be hypothesis generating and descriptive in nature. Descriptive statistics will be summarized and the blood and tissue marker data will be correlated with clinical endpoints (response, DCR12, duration of response, OS, PFS, adverse events, etc.). For time-to-event data, the Kaplan-Meier method will be used. For categorical data, will use the Fisher's exact test. For marker data used to predict binary outcomes (i.e. response vs. no response), will use logistic regression models.
Time Frame: Baseline up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Mechanisms of Resistance in ctDNA Profile After Therapy With a PARPi and a PD-1 Inhibitor
Description: as for outcome 9
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Tumor Microenvironment for Immune Related Changes (Immune Infiltration, PD-L1 and PD-1 Expression, Tumor-infiltrating Lymphocytes)
Description: as for outcome 9
Time Frame: Up to 5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Genetic Profile of the Tumor Pre- and Post-treatment
Description: as for outcome 9
Time Frame: Baseline up to 5 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Changes in the Cytokine Profile Pre- and Post-treatment
Description: as for outcome 9
Time Frame: Baseline up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 years and 5 months
Arm/Group | Treatment (Niraparib, Dostarlimab)
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Niraparib, Dostarlimab) (N=20)
Asystole (Cardiac disorders) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Niraparib, Dostarlimab) (N=20)
Anemia (Blood and lymphatic system disorders) | 19 (59)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (11)
Abdominal distension (Gastrointestinal disorders) | 1 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Ascites (Gastrointestinal disorders) | 1 (6)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 17 (52)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Pain (General disorders) | 13 (42)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (5)
Anorectal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (6)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 6 (9)
Blood bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 5 (19)
Lymphocyte count decreased (Investigations) | 5 (13)
Neutrophil count decreased (Investigations) | 2 (4)
Platelet count decreased (Investigations) | 8 (20)
Weight loss (Investigations) | 1 (3)
White blood cell decreased (Investigations) | 2 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (21)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (4)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3)
Hypertension (Vascular disorders) | 1 (5)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT04493060/Prot_SAP_002.pdf
  • Informed Consent Form (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT04493060/ICF_001.pdf